CLINICAL TRIAL: NCT02880644
Title: Ultra-wide Fluorescein angiograpHy to Evaluate the Progression of Retinal ischeMia After aflibErcept Injections in patientS With Central Retinal Vein Occlusion in Real Life (HERMES Study)
Brief Title: Ultra-wide Fluorescein Angiography in Patients With Central Retinal Vein Occlusion Treated by Afilbercept
Acronym: HERMES
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Collaborators: Bayer (Industry); Association Clinique Thérapeutique Infantile du val de Marne (Other)
Responsible Party: Principal Investigator, Agnes Glacet-Bernard, Ophtalmologist, Centre Hospitalier Intercommunal Creteil
Other Study IDs: HERMES
Record Dates: First submitted 2016-08-23; First posted 2016-08-26 (Estimated); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Retinal Vein Occlusion
Keywords: Central retinal vein occlusion; OCT-A; CRVO
MeSH Terms: conditions — Retinal Vein Occlusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: Yes

SUMMARY:
In patients with macular edema secondary to CRVO, Aflibercept demonstrated efficacy and safety in 2 parallel trials, interventional phase III studies, COPERNICUS study performed in United States and GALILEO study performed in Europe and Asia/Pacific.

With the project of Hermes Study, the first observational study conducted in France in patients with CRVO and treated with aflibercept, we would like to evaluate in real life the monitoring and the use of Aflibercept. The primary objective of this study will also be based on anatomic outcomes. The evolution of retinal ischemia and the degree of non-retinal perfusion will be particularly evaluated by using ultra wide field angiography technology.

DETAILED DESCRIPTION:
The pathophysiology of Central Retinal Vein Occlusion (CRVO) is incompletely understood, but a significant slow-down in blood flow, caused by various predisposing factors, results in the release of VEGF, leading to the breakdown of the blood-retinal-barrier and finally to macular edema. The level of VEGF has been also correlated with neovascularization and vascular permeability in patients with ischemic CRVO. Several treatments have been used to treat patients with CRVO such as hemodilution, surgery, laser treatment and corticoids injection. However anti-vascular endothelial growth factor (anti-VEGF) agents administered by intravitreal injection, improve both visual and anatomic outcomes in patients with macular edema secondary to CRVO. Aflibercept is a fusion protein, use by intravitreal injection. In patients with macular edema secondary to CRVO, Aflibercept demonstrated efficacy and safety in 2 parallel trials, interventional phase III studies, COPERNICUS study performed in United States and GALILEO study performed in Europe and Asia/Pacific. In these studies, anatomic outcomes such as ischemic progression and retinal perfusion status were evaluated as secondary objectives; the primary objective of these studies was visual outcome.

With the project of Hermes Study, the first observational study conducted in France in patients with CRVO and treated with aflibercept, we would like to evaluate in real life the monitoring and the use of Aflibercept. The primary objective of this study will also be based on anatomic outcomes. The evolution of retinal ischemia and the degree of non-retinal perfusion will be particularly evaluated by using ultra wide field angiography technology.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman aged 18 years or more
* Patients with a diagnosis of CRVO (presence of retinal hemorrhages associated with vein dilation and tortuosity in the 4 quadrants)
* The decision for treatment with Aflibercept (Eylea®) has been made for patients with a decrease in Best Corrected Visual Acuity (BCVA) and macular edema
* Duration of CRVO not more than 4 months
* Naïve patients. Patient with previous CRVO (more than 12 months before the inclusion date) which completely resolved (normalization of visual acuity and fundus examination) and who experienced a recurrence of CRVO are also considered naive
* Patient who agrees to participate to the study and who has given his/her written, informed consent

Exclusion Criteria:

* Patient with another retinal disease in the study eye: diabetic retinopathy, maculopathy of any cause (age-related macular degeneration, epimacular membrane, myopia, etc) responsible for decreased vision, advanced glaucoma, cataract severely affecting vision and/or requiring surgical treatment during the 24 months study period
* Patient who does not meet the local indication criteria for aflibercept treatment. Contraindications listed in the SmPCs must be taken into account including:
* Hypersensitivity to the active substance aflibercept or to any of the excipients listed in SmPC of the product
* Active or suspected ocular or periocular infection
* Active severe intraocular inflammation
* CRVO complicated with neovascularization of the anterior segment
* Patient who has previously undergone laser panretinal photocoagulation, grid-laser or photodynamic therapy, any anti-VEGF or corticoids intravitreal injections in the study eye
* Patient already included in the study for the treatment of the fellow eye
* Pregnant or breastfeeding woman
* Lack of effective contraception for women of childbearing age
* Patient taking part in an interventional study
* Patients not covered by the French Health Insurance

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with central retinal vein occlusion
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2017-01-26 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in non-perfused areas in both macula and peripheral retina at 12 months | Baseline and 12 months

SECONDARY OUTCOMES:
Change in visual acuity from baseline to months 3, 6, 12 and 24 | Baseline and 3, 6, 12 and 24 months
Change from baseline in non-perfused areas in both macula and peripheral retina at 3, 6 and 12 months | Baseline and 3, 6 and 12 months
Mean time between the last two injections | Up to 18 weeks
Mean number of injections by patient from baseline to end-of-study visit | From baseline to 24 months
Mean number of visits by patient from baseline to end-of-study visit | From baseline to 24 months
Change from baseline in central retinal thickness at 3, 6, 12 and 24 months | Baseline and 3, 6, 12 and 24 months
Change in vascular density in OCT-A from baseline to months 3, 6, 12, 24 | Baseline and 3, 6, 12 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Agnès GLACET-BERNARD, MD, Principal Investigator — Centre Hospitalier Intercommunal Créteil
Locations (9):
- France (9):
  - Centre Hospitalier Intercommunal Créteil, Créteil
  - Centre Monticelli Paradis d'Ophtalmologie, Marseille
  - Centre Hospitalier Universitaire De Nantes, Nantes
  - CHU Nice-Saint-Roch, Nice
  - Centre d'exploration ophtalmologique de l'odéon, Paris
  - Centre d'Imagerie et de laser, Paris
  - CHNO des Quinze-Vingts, Paris
  - Hôpital Lariboisière - APHP, Paris
  - Hôpital Robert Debré - CHU Reims, Reims

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Williamson TH. Central retinal vein occlusion: what's the story? Br J Ophthalmol. 1997 Aug;81(8):698-704. doi: 10.1136/bjo.81.8.698. No abstract available. PMID 9349161
- [Background] Hayreh SS. So-called "central retinal vein occlusion". I. Pathogenesis, terminology, clinical features. Ophthalmologica. 1976;172(1):1-13. doi: 10.1159/000307579. PMID 1250571
- [Background] Fujikawa M, Sawada O, Miyake T, Kakinoki M, Sawada T, Kawamura H, Ohji M. Correlation between vascular endothelial growth factor and nonperfused areas in macular edema secondary to branch retinal vein occlusion. Clin Ophthalmol. 2013;7:1497-501. doi: 10.2147/OPTH.S46817. Epub 2013 Jul 19. PMID 23901258
- [Background] Noma H, Minamoto A, Funatsu H, Tsukamoto H, Nakano K, Yamashita H, Mishima HK. Intravitreal levels of vascular endothelial growth factor and interleukin-6 are correlated with macular edema in branch retinal vein occlusion. Graefes Arch Clin Exp Ophthalmol. 2006 Mar;244(3):309-15. doi: 10.1007/s00417-004-1087-4. Epub 2005 Aug 13. PMID 16133018
- [Background] Natural history and clinical management of central retinal vein occlusion. The Central Vein Occlusion Study Group. Arch Ophthalmol. 1997 Apr;115(4):486-91. doi: 10.1001/archopht.1997.01100150488006. PMID 9109757
- [Background] Evaluation of grid pattern photocoagulation for macular edema in central vein occlusion. The Central Vein Occlusion Study Group M report. Ophthalmology. 1995 Oct;102(10):1425-33. doi: 10.1016/s0161-6420(95)30849-4. PMID 9097788
- [Background] Opremcak EM, Rehmar AJ, Ridenour CD, Kurz DE. Radial optic neurotomy for central retinal vein occlusion: 117 consecutive cases. Retina. 2006 Mar;26(3):297-305. doi: 10.1097/00006982-200603000-00008. PMID 16508430
- [Background] Glacet-Bernard A, Atassi M, Fardeau C, Romanet JP, Tonini M, Conrath J, Denis P, Mauget-Faysse M, Coscas G, Soubrane G, Souied E. Hemodilution therapy using automated erythrocytapheresis in central retinal vein occlusion: results of a multicenter randomized controlled study. Graefes Arch Clin Exp Ophthalmol. 2011 Apr;249(4):505-12. doi: 10.1007/s00417-010-1532-5. Epub 2010 Oct 17. PMID 20953877
- [Background] Ip MS, Scott IU, VanVeldhuisen PC, Oden NL, Blodi BA, Fisher M, Singerman LJ, Tolentino M, Chan CK, Gonzalez VH; SCORE Study Research Group. A randomized trial comparing the efficacy and safety of intravitreal triamcinolone with observation to treat vision loss associated with macular edema secondary to central retinal vein occlusion: the Standard Care vs Corticosteroid for Retinal Vein Occlusion (SCORE) study report 5. Arch Ophthalmol. 2009 Sep;127(9):1101-14. doi: 10.1001/archophthalmol.2009.234. PMID 19752419
- [Background] Haller JA, Bandello F, Belfort R Jr, Blumenkranz MS, Gillies M, Heier J, Loewenstein A, Yoon YH, Jacques ML, Jiao J, Li XY, Whitcup SM; OZURDEX GENEVA Study Group. Randomized, sham-controlled trial of dexamethasone intravitreal implant in patients with macular edema due to retinal vein occlusion. Ophthalmology. 2010 Jun;117(6):1134-1146.e3. doi: 10.1016/j.ophtha.2010.03.032. Epub 2010 Apr 24. PMID 20417567
- [Background] Campochiaro PA, Brown DM, Awh CC, Lee SY, Gray S, Saroj N, Murahashi WY, Rubio RG. Sustained benefits from ranibizumab for macular edema following central retinal vein occlusion: twelve-month outcomes of a phase III study. Ophthalmology. 2011 Oct;118(10):2041-9. doi: 10.1016/j.ophtha.2011.02.038. Epub 2011 Jun 29. PMID 21715011
- [Background] Heier JS, Clark WL, Boyer DS, Brown DM, Vitti R, Berliner AJ, Kazmi H, Ma Y, Stemper B, Zeitz O, Sandbrink R, Haller JA. Intravitreal aflibercept injection for macular edema due to central retinal vein occlusion: two-year results from the COPERNICUS study. Ophthalmology. 2014 Jul;121(7):1414-1420.e1. doi: 10.1016/j.ophtha.2014.01.027. Epub 2014 Mar 27. PMID 24679444
- [Background] Ogura Y, Roider J, Korobelnik JF, Holz FG, Simader C, Schmidt-Erfurth U, Vitti R, Berliner AJ, Hiemeyer F, Stemper B, Zeitz O, Sandbrink R; GALILEO Study Group. Intravitreal aflibercept for macular edema secondary to central retinal vein occlusion: 18-month results of the phase 3 GALILEO study. Am J Ophthalmol. 2014 Nov;158(5):1032-8. doi: 10.1016/j.ajo.2014.07.027. Epub 2014 Jul 25. PMID 25068637